CLINICAL TRIAL: NCT00761878
Title: Evaluation of the PlasmaJet Neutral Argon Plasma System for Skin Regeneration and Comparison With the Rhytec Portrait PSR Plasma System
Brief Title: Evaluation of the PlasmaJet Neutral Argon Plasma System to Treat Skin Ageing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Plasma Surgical Inc (Industry)
Responsible Party: Dr Denis F Branson, Denis F Branson MD
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSI-2007-07
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-07

CONDITIONS: Skin Aging
Keywords: Skin aging; Skin wrinkling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Skin treatment (Active Comparator)
  Interventions: Procedure: Exposure to plasma energy

INTERVENTIONS:
Procedure: Exposure to plasma energy — Non-invasive exposure to pulsed plasma to the unbroken skin over half of the facial area

SUMMARY:
The purpose of this study is to determine the comparative effects of the PlasmaJet neutral argon plasma system and the Rhytec Portrait PRS nitrogen plasma system in the treatment of aging facial skin

ELIGIBILITY:
Inclusion Criteria:

* request for treatment to improve facial skin

Exclusion Criteria:

* pregnancy
* history of HIV infection
* autoimmune or connective tissue disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Assessment of skin appearance and condition by photography and digital image analysis | At intervals for up to 12 months

SECONDARY OUTCOMES:
Assessment of skin condition and dermal architecture by ultrasound imaging | At intervals for up to 12 months
Assessment of skin elasticity by non-invasive means | At intervals for up to 12 months
Assessment of pain during treatment | During treatment

CONTACTS AND LOCATIONS:
Overall Officials: Denis F Branson, MD, Principal Investigator — Denis F Branson MD
Locations (1):
- Denis F Branson MD, Fayetteville, New York, United States